CLINICAL TRIAL: NCT02538302
Title: Minirin Versus Oxybutynin for Nocturnal Enuresis in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Principal Investigator, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 92.121.505
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Nocturnal Enuresis
Keywords: Minirin; Oxybutynin; Nocturnal enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minirin (Experimental): 120 microgram per day for 2 months, then 60 microgram per day for 2 months, then 60 microgram every two days for two months
  Interventions: Drug: Minirin
- Oxybutynin (Active Comparator): 5 mg Oxybutynin twice a daily for 6 months
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Minirin — Minirin 5 to 10 mg daily for 6 months
  Other Names: Desmopressin acetate
  Arms: Minirin
Drug: Oxybutynin — Oxybutynin 5 to 10 mg daily for 6 months
  Other Names: Ditropan
  Arms: Oxybutynin

SUMMARY:
Nocturnal enuresis is among the most common disorders in children. The aim of current study was to compare the efficacy and safety of Minirin and oxybutynin for treatment of nocturnal enuresis in children in Bandar Abbas in 2014.

DETAILED DESCRIPTION:
Nocturnal enuresis is among the most common disorders in children. Several pharmacological and non-pharmacological treatments are available for nocturnal enuresis. Studies for reaching the best pharmacological treatment for this disorder are continuing. The aim of current study was to compare the efficacy and safety of Minirin and oxybutynin for treatment of nocturnal enuresis in children in Bandar Abbas in 2014.

ELIGIBILITY:
Inclusion Criteria:

* >5 years old
* Nocturnal enuresis
* Candidate for pharmacological treatment

Exclusion Criteria:

* Children who their parents did noted filled the informed consent form
* Impossibility of follow up during the study period
* History of seizure
* History of rheumatologic disorders such as sjogren's disease

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ّFrequency of nocturnal enuresis | 6 months
  Number of participants with nocturnal enuresis

SECONDARY OUTCOMES:
Frequency of urinary incontinency | 6 months
  Number of participants with urinary incontinency
Frequency of urgency | 6 months
  Number of participants with urgency
Frequency of Xerostomia | 6 months
  Number of participants with Xerostomia
Frequency of Xerophthalmia | 6 months
  Number of participants with Xerophthalmia
Frequency of Blurred vision | 6 months
  Number of participants with Blurred vision
Frequency of Dysphagia | 6 months
  Number of participants with Dysphagia
Frequency of constipation | 6 months
  Number of participants with constipation
Frequency of Diarrhea | 6 months
  Number of participants with Diarrhea
Frequency of Headache | 6 months
  Number of participants with Headache
Frequency of Seizure | 6 months
  Number of participants with Seizure
Frequency of Epistaxis | 6 months
  Number of participants with Epistaxis
Frequency of Abdominal pain | 6 months
  Number of participants with Abdominal pain
Frequency of Vomiting | 6 months
  Number of participants with Vomiting
Frequency of Ear ache | 6 months
  Number of participants with Ear ache
Frequency of Rhinitis | 6 months
  Number of participants with Rhinitis
Frequency of Chest pain | 6 months
  Number of participants with Chest pain
Frequency of Increase in appetite | 6 months
  Number of participants with Increase in appetite

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Mahboobi, M.D, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Shahid Mohammadi hospital, Bandar Abbas, Hormozgan, Iran

REFERENCES:
- [Derived] Ghasemi K, Esteghamati M, Mohammadzadeh M, Zare S. Desmopressin versus Oxybutynin for Nocturnal Enuresis in Children in Bandar Abbas: A Randomized Clinical Trial. Electron Physician. 2016 Mar 25;8(3):2187-93. doi: 10.19082/2187. eCollection 2016 Mar. PMID 27123229